CLINICAL TRIAL: NCT04597541
Title: A Phase I/II Trial of AK112 in Advanced Solid Tumor
Brief Title: A Study of AK112 for Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK112-102
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): AK112
  Interventions: Drug: AK112

INTERVENTIONS:
Drug: AK112 — AK112 is a PD1/VEGF bispecific antibody;AK112 is given by intravenous infusion.

SUMMARY:
This study is to characterize the safety, tolerability, pharmacokinetics (PK), immunogenicity, pharmacodynamics (PD) and anti-tumor activity of AK112, a PD-1/VEGF bispecific antibody, as a single agent in adult subjects with advanced solid tumor malignancies. This trial is a two parts, phase I/II study. All patients are advanced solid tumor, Eastern Cooperative Oncology Group (ECOG) performance status 0-1. Part one is dose escalation phase,part two is dose expansion phase. The primary end point is safety. Secondary end points are objective response rate,progression-free survival and overall survival per RECIST1.1.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years old (at the time consent is obtained);
* Be able and willing to provide written informed consent and to comply with all requirements of study participation (including all study procedures);
* Have histologically- or cytologically-confirmed diagnosis of advanced solid tumor;
* Available archived tumor tissue sample to allow for correlative biomarker studies. In the setting where archival material is unavailable or unsuitable for use, the subject must consent and undergo fresh tumor biopsy;
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or
* Subject must have at least one measurable lesion according to RECIST Version1.1;
* Adequate organ function;
* Females of childbearing potential and non-sterilized males who are sexually active must use an effective method;
* Adequate life expectancy.

Exclusion Criteria:

* History of severe hypersensitivity reactions to other mAbs;
* Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5.0 Grade 0 or 1, or to levels dictated in the inclusion/exclusion criteria;
* Major surgical procedure within 30 days prior to the first dose of AK112 or still recovering from prior surgery;
* Receipt of any immunotherapy, any conventional or investigational systemic anticancer therapy within 4 weeks prior to the first dose of AK112 except for treatment with small-molecule tyrosine kinase-targeted agents within 2 weeks prior to the first dose of AK112;
* History of primary immunodeficiency;
* Active or prior documented inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis);
* History of organ transplant or hematopoietic stem cell that requires use of immunosuppressives;
* Known allergy or reaction to any component of the AK112 formulation;
* History of interstitial lung disease or non-infectious pneumonitis except for those induced by radiation therapies;
* Known history of tuberculosis;
* Known history of HIV;
* Receipt of live attenuated vaccination within 30 days prior to the first dose of AK112;
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | From time ICF is signed until 90 days after last dose of AK112
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product.
  temporally associated with the use of study treatment, whether or not considered related to the study treatment
Number of participants with DLTs | During the first four weeks of treatment
  DLTs will be assessed during the first 4 weeks of treatment for dose-escalation phase and are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug, and unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first cycle (4 weeks) of treatment.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD at 16 and 24 weeks respectively) based on RECIST Version 1.1.
Progression-free survival (PFS) | Up to 2 years
  Progression-free survival is defined as the time from the start of treatment with AK112 until the first documentation of disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 2 years
  Overall survival is defined as the time from the start of treatment with AK112 until death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Wang F, Wei X, Zheng Y, Wang J, Ying J, Chen X, Luo S, Luo H, Yu X, Chen B, Ma L, Xu R. Safety, Pharmacokinetics, and Pharmacodynamics Evaluation of Ivonescimab, a Novel Bispecific Antibody Targeting PD-1 and VEGF, in Chinese Patients With Advanced Solid Tumors. Cancer Med. 2025 Mar;14(6):e70653. doi: 10.1002/cam4.70653. PMID 40114411